CLINICAL TRIAL: NCT04741672
Title: Home Support for Mothers Whose Premature Infants Discharged From the Neonatal Intensive Care Unit: A Randomized Controlled Study
Brief Title: Home Support for Mothers Whose Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Arzu Akcan, Assistant Professor, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 19113
Record Dates: First submitted 2021-01-25; First posted 2021-02-05 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Infant, Premature, Diseases; Mothers
Keywords: Infant; Mothers
MeSH Terms: conditions — Infant, Premature, Diseases

STUDY DESIGN:
Intervention Model Description: This was pretest-posttest design, randomized controlled trial.
Who Masked: Participant
Masking Description: The control and intervention group will be formed by randomization. The intervention and control group will be defined as group 1 and group 2 for statistical analysis. Data analysis will be evaluated and reported by the statistician. Also the statistician will be blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Providing guidance and calling after discharge routine procedure.
  Interventions: Behavioral: Providing guidance after discharge routine procedure and calling one week after discharge.; Behavioral: Discharge routine procedure.
- Control group (Experimental): Discharge routine procedure.
  Interventions: Behavioral: Discharge routine procedure.

INTERVENTIONS:
Behavioral: Providing guidance after discharge routine procedure and calling one week after discharge. — Guidance will be given to mothers after routine discharge. After one week, she will be called by phone and her questions about infant care will be answered.
  Arms: Intervention group
Behavioral: Discharge routine procedure. — Discharge routine procedure.

SUMMARY:
Premature births are a challenging process for parents in many ways. Especially after the treatment and care in the hospital, they are concerned about whether they will be able to provide adequate care for their baby at home. The aim of this study is to examine the effect of the guide and telephone support given to mothers whose premature infants were discharged from the neonatal intensive care unit on the perceived maternal self-efficacy and state anxiety levels.

DETAILED DESCRIPTION:
The study was planned as a randomized controlled trial with a single blind, pretest-posttest design. This study will be conducted between February 2021 and March 2022 with premature infants mothers. The sample of the study will be mothers (n = 102) of premature infants discharged from Antalya Training and Research Hospital Neonatal Intensive Care Unit. 51 mothers participating in the study will be given a premature infant home care guide after the discharge routine procedures are completed. In addition, mothers will be given an appointment for a phone call a week later. No intervention will be applied to the other 51 mothers after their discharge routine. Data will be collected by Mother-Infant Descriptive Information Form, Perceived Maternity Self-Efficacy Scale (PMSES), State Anxiety Inventory (SAI). Data will be collected with forms and scales immediately after discharge (pre-test) and in the 4th week after discharge (post-test). Ethics Committee and Institutional Permission was obtained for the study. In addition, written consent will be obtained from the participants. Statistical analysis will be done using SPSS 23.0 and significance will be evaluated at p <0.05. Support will be received in the analysis phase of the Statistical Information Unit of Akdeniz University. It is predicted that the new information obtained from the research data will guide the education of premature infant mothers and new researches.

ELIGIBILITY:
Inclusion Criteria:

* The infant was born prematurely (37 weeks of gestation + 6 days earlier),
* Does not have advanced congenital anomalies in the baby,
* Who will carry out the primary care of the infant at home,
* Reading and writing,
* Can speak and understand Turkish,
* Mothers who agreed to participate in the study

Exclusion Criteria:

* Incomplete filling of the forms
* Mothers who previously had training in newborn care

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Perceived Maternity Self-Efficacy Scale | 0-1 months (Immediately before discharge training and 4 weeks after discharge training completion)
  The scale, valid and reliable in our country by Kadiroglu (2018), has 19 items and three sub-dimensions.A minimum of 19 and a maximum of 76 points can be obtained on the scale.
State Anxiety Inventory | 0-1 months (Immediately before discharge training and 4 weeks after discharge training completion)
  The scale was developed to measure what has been felt for the last 7 days. It is a Likert-type scale consisting of 20 items and graded between 1 and 4. The scores obtained from the scale range from 20 to 80.

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Akcan, PhD, Study Director — Akdeniz Universtiy; Ezgi Boz, Postgraduate, Study Chair — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee SY, Chau JPC, Choi KC, Lo SHS. Feasibility of a guided participation discharge program for very preterm infants in a neonatal intensive care unit: a randomized controlled trial. BMC Pediatr. 2019 Nov 4;19(1):402. doi: 10.1186/s12887-019-1794-y. PMID 31684903